CLINICAL TRIAL: NCT02205424
Title: Is Stroke Neurodegenerative? A Longitudinal Study of Brain Volume and Cognitive Decline Following Stroke (CANVAS: Cognition And Neocortical Volume After Stroke).
Brief Title: Cognition And Neocortical Volume After Stroke
Acronym: CANVAS
Status: Completed | Type: Observational
Sponsor: The Florey Institute of Neuroscience and Mental Health (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Amy Brodtmann, Prof Amy Brodtmann, The Florey Institute of Neuroscience and Mental Health
Other Study IDs: APP-1020526
Record Dates: First submitted 2014-03-20; First posted 2014-07-31 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Ischaemic Stroke; Alzheimer's Disease; Vascular Dementia
Keywords: Ischaemic stroke; Alzheimer's disease; Brain volume; Cortical thickness; Magnetic Resonance Imaging
MeSH Terms: conditions — Ischemic Stroke; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood for APOE estimation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ischaemic stroke patients: Patients who have suffered an ischaemic stroke, as determined clinically and verified with imaging (CT brain; MRI).
- Healthy control participants: People who have never suffered a stroke, and are matched to the ischaemic stroke patient group according to age, education, and vascular risk factors.

SUMMARY:
Stroke and dementia are two of the most common and disabling conditions worldwide, responsible for an enormous and growing burden of disease. There is increasing awareness that the two conditions are linked, with cognitive impairment and dementia common after stroke, vascular dementia accounting for about one-fifth of all dementia cases and recent evidence on the contribution of vascular risk factors to Alzheimer's disease. Yet little is known about whether brain volume loss - a hallmark of dementia - occurs after stroke, and whether such atrophy is related to cognitive decline. The aim of this research is to establish whether stroke patients have reductions in brain volume in the first three years post-stroke compared to control subjects, and whether regional and global brain volume change is associated with post-stroke dementia in order to elucidate potential causal mechanisms (including genetic markers, amyloid deposition and vascular risk factors). The hypotheses are that stroke patients will exhibit greater brain volume loss than comparable cohorts of stroke-free controls, and further, that stroke patients who develop dementia will exhibit greater global and regional brain volume loss than those who do not dement. An understanding of whether stroke is neurodegenerative, and in which patients, may be used to help guide the early delivery of disease-modifying therapies.

DETAILED DESCRIPTION:
Our primary outcome measure was total brain volume (TBV) change between the 3-month and 3-year time-points compared between stroke patients and controls.

Secondary outcome 1 was TBV change between 3-months and 3-years comparing CN and CI stroke participants. TBV at 3-months will be adjusted for CCI scores, and years of education; the latter as it is correlated with cognitive performance and post-stroke dementia risk, but not for stroke lesion volume as no conclusive evidence for an effect has been demonstrated previously.

Secondary outcome 2 was hippocampal volume (HV) change between 3-months and 3-years in stroke patients and controls with adjustments identical to primary outcome.

Secondary outcome 3 was the comparison of HV change between 3-months and 3-years comparing CN and CI stroke participants with adjustments identical to secondary outcome 1.

See published protocol and uploaded statistical analysis plan for detailed description.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stroke
2. Aged greater than 18 years;
3. Able to have cognitive testing and MRI scan; and
4. Able to give informed consent

Exclusion Criteria:

1. Significant medical comorbidities precluding participation in cognitive testing, or making survival for three years unlikely;
2. Normal exclusion criteria for MRI; e.g., implanted metal, severe claustrophobia;
3. Pre-existing dementia
4. Pregnancy, as a precaution to prevent exposing them to multiple MRI scans in a 12-month period
5. People in existing dependent or unequal relationships with any member of the research team, to protect against coercion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ischaemic stroke patients will have been admitted to the Acute Neurology Units of the Austin Hospital (Heidelberg), Royal Melbourne Hospital (Parkville), and Box Hill Hospital (Box Hill).
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in total brain volume between 3 month and 3 year time-points | Between 3 months and 3 years post-stroke
  We will examine changes in brain volume between the 3 month and 3 year time-points in ischemic stroke patients and healthy age-matched control participants

SECONDARY OUTCOMES:
Comparison of total brain volume (TBV) change between 3 month and 3 year time-points in those who were cognitively normal (CN) versus cognitively impaired (CI) determined at the 3 months post-stroke time point. | Between 3 months and 3 years post-stroke
  Secondary outcome 1 was TBV change between 3-months and 3-years comparing CN and CI stroke participants.
Difference in hippocampal volume between 3 month and 3 year time-points in stroke and control participants. | Between 3 months and 3 years post-stroke
  Secondary outcome 2 was hippocampal volume (HV) change between 3-months and 3-years in stroke patients and controls with adjustments identical to primary outcome.
Comparison of hippocampal volume change between 3 month and 3 year time-points in those who were cognitively normal versus cognitively impaired at 3 months post-stroke. | Between 3 months and 3 years post-stroke
  Secondary outcome 3 was the comparison of HV change between 3-months and 3-years comparing CN and CI stroke participants with adjustments identical to secondary outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Amy G Brodtmann, MBBS PhD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health
Locations (3):
- Australia (3):
  - Eastern Health, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Melbourne Health, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egorova-Brumley N, Dhollander T, Khan W, Khlif MS, Ebaid D, Brodtmann A. Changes in White Matter Microstructure Over 3 Years in People With and Without Stroke. Neurology. 2023 Apr 18;100(16):e1664-e1672. doi: 10.1212/WNL.0000000000207065. Epub 2023 Feb 15. PMID 36792378
- [Derived] Hung SH, Khlif MS, Kramer S, Werden E, Bird LJ, Campbell BCV, Brodtmann A. Poststroke White Matter Hyperintensities and Physical Activity: A CANVAS Study Exploratory Analysis. Med Sci Sports Exerc. 2022 Sep 1;54(9):1401-1409. doi: 10.1249/MSS.0000000000002946. Epub 2022 Apr 25. PMID 35482768
- [Derived] Brodtmann A, Werden E, Khlif MS, Bird LJ, Egorova N, Veldsman M, Pardoe H, Jackson G, Bradshaw J, Darby D, Cumming T, Churilov L, Donnan G. Neurodegeneration Over 3 Years Following Ischaemic Stroke: Findings From the Cognition and Neocortical Volume After Stroke Study. Front Neurol. 2021 Oct 22;12:754204. doi: 10.3389/fneur.2021.754204. eCollection 2021. PMID 34744989
- [Derived] Brodtmann A, Khlif MS, Egorova N, Veldsman M, Bird LJ, Werden E. Dynamic Regional Brain Atrophy Rates in the First Year After Ischemic Stroke. Stroke. 2020 Sep;51(9):e183-e192. doi: 10.1161/STROKEAHA.120.030256. Epub 2020 Aug 10. PMID 32772680
- See also: Primary and secondary hypotheses reporting — https://www.medrxiv.org/content/10.1101/2021.08.03.21261461v1